CLINICAL TRIAL: NCT03252431
Title: A Phase III, Randomized, Multi-Centre, Open-Label, Fixed Dose, Neulasta® Active-Controlled Clinical Trial of F-627 in Women With Breast Cancer Receiving Myelotoxic Chemotherapy
Brief Title: Neulasta-controlled Trial of F-627 in Women With Breast Cancer Receiving Myelotoxic Chemotherapy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EVIVE Biotechnology (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GC-627-05
Record Dates: First submitted 2017-08-14; First posted 2017-08-17 (Actual); Results first posted 2021-05-07 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2021-04

CONDITIONS: Breast Cancer; Neutropenia
MeSH Terms: conditions — Breast Neoplasms; Neutropenia | interventions — pegfilgrastim

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- F-627 (Experimental): F-627, 20 mg fixed dose pre-filled syringe, administered on Day 2 of each of 4 chemotherapy cycles.
  Interventions: Drug: F-627
- Neulasta (Active Comparator): 6 mg fixed dose Neulasta®, administered on Day 2 of each of 4 chemotherapy cycles
  Interventions: Drug: Neulasta

INTERVENTIONS:
Drug: F-627 — single dose pre-filled syringe
  Arms: F-627
Drug: Neulasta — single dose pre-filled syringe
  Other Names: pegfilgrastim
  Arms: Neulasta

SUMMARY:
This is a randomized, multi-center, single dose, open-label and Neulasta controlled phase 3 study to evaluate the efficacy and safety of F-627 in women with Stage I - III invasive breast cancer receiving chemotherapy treatment.

DETAILED DESCRIPTION:
This is a Phase III, global, two arm, open label clinical study will randomize approximately 400 female subjects (approximately 200 per arm) with Stage I - III invasive breast cancer who are to receive neoadjuvant or adjuvant myelotoxic TC chemotherapy treatment (docetaxel + cyclophosphamide, 75 and 600 mg/m2, respectively). Subjects in this study will be those who are scheduled to undergo at least four 21-day cycles of chemotherapy treatment. Subjects may be scheduled for more than 4 cycles of chemotherapy; however, study participation will be limited to a subject's first 4 cycles.

The primary objective of this study will be to evaluate the efficacy of F-627 given as a single fixed dose (20 mg) pre-filled syringe as compared to Neulasta® standard dosing (6 mg) in the first chemotherapy cycle. The primary endpoint will be the duration of grade 4 (severe) neutropenia - the number of days in which the patient has had an absolute neutrophil count (ANC <0.5 x 10^9/L) observed in chemotherapy cycle 1.

Approximately 24 hours after chemotherapy completion in each cycle (Day 2 of the cycle), subjects will receive one of the following treatments:

Arm 1: F-627, 20 mg fixed dose pre-filled syringe, administered on Day 2 of each of 4 chemotherapy cycles.

Arm 2: 6 mg fixed dose Neulasta®, administered on Day 2 of each of 4 chemotherapy cycles Randomization will occur in an equal ratio (1:1) using a central randomization system (IWRS) on Day 1 of the study, the day of chemotherapy administration for the first chemotherapy cycle.

This study is open-label, however, study drug injections are to be administered separately by qualified study personnel to allow study investigators to remain blinded and perform study assessments without knowledge of treatment assignment.

ELIGIBILITY:
Inclusion Criteria:

1. Show evidence of a personally signed and dated informed consent document indicating that the patient has been informed of all pertinent aspects of the trial.
2. Females ≥18 years of age.
3. Diagnosed with Stage I-III breast cancer.
4. Subject is scheduled to undergo 4 cycles of neoadjuvant or adjuvant TC chemotherapy (docetaxel, cyclophosphamide, 75, 600 mg/m2, respectively).
5. ECOG Performance status of ≤2.
6. WBC count ≥4.0 × 109/L, hemoglobin ≥11.5 g/dL and a platelet count ≥150 × 109/L.
7. Demonstrate adequate renal, hepatic, and cardiac function (liver function tests [alanine aminotransferase {ALT}, aspartate aminotransferase {AST}, alkaline phosphatase, and total bilirubin]) should be less than 2.5x the upper limits of normal (ULN). Serum creatinine should be less than 1.7x ULN.
8. All subjects must agree to use at least one of the following types of contraception: intrauterine device, implantable progesterone device, progesterone intramuscular injection, or oral contraceptive, which has been started at least one month prior to visit one and will continue for the duration of the trial. The contraceptive patch or condom use with spermicide is also acceptable forms of contraception as long as they will be used continually throughout the duration of the trial.

Exclusion Criteria:

1. Subject is <18 years of age.
2. Disease progression has occurred while receiving a taxane regimen.
3. Subject has undergone radiation therapy within 4 weeks of enrollment.
4. Subject has undergone bone marrow or stem-cell transplantation.
5. Subject has a history of prior malignancy other than breast cancer that is NOT in remission.
6. Subjects that have used G-CSF or any other drug that may potentiate the release of neutrophils (i.e., lithium) within 6 weeks of the screening period are excluded.
7. Subject has had chemotherapy within 180 days of screening.
8. Subject has documented congestive heart failure, cardiomyopathy or myocardial infarction by clinical diagnosis, electrocardiogram (ECG) test, or any other relevant test.
9. History of alcohol or drug abuse that would interfere with the ability to be compliant with the study procedure.
10. Unwillingness to participate in the study.
11. Any underlying medical condition that, in the Investigator's opinion, would make the administration of study drug hazardous to the patient or that would obscure the interpretation of adverse events.
12. Receiving other investigational drugs or biologics within 1 month or five half lives of enrollment (if known), which ever is less.
13. Any condition, which can cause splenomegaly.
14. Chronic constipation or diarrhea, irritable bowel syndrome, inflammatory bowel disease.
15. ALT, AST, alkaline phosphatase, total bilirubin ≥2.5x ULN.
16. Subject with active infection, or known to be infected with chronic active Hepatitis B within the last 1 year (unless shown at the time of study entry to be Hepatitis B antigen negative), or having any history of Hepatitis C.
17. Women who are pregnant or breast-feeding.
18. Subject known to be seropositive for HIV, or who have had an AIDS defining illness or a known immunodeficiency disorder.
19. Subject with a history of tuberculosis or exposure to tuberculosis. Patients that have received a prior chest X-ray for suspicion of tuberculosis are also excluded unless they have been confirmed to be PPD negative or they had latent tuberculosis that has been previously treated.
20. Subjects with Sickle Cell disease
21. Subjects with known hypersensitivity to E.coli derived proteins' pegfilgrastim' filgrastim, or any other component of the study drug.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2020-03-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Glaspy, MD, Principal Investigator — University of California at Los Angeles
Locations (1):
- University of California Los Angeles (UCLA) - Jonsson Comprehensive Cancer Center (JCCC), Los Angeles, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | F-627 | Neulasta
Started | 197 | 196
Completed | 186 | 187
Not Completed | 11 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | F-627 | Neulasta | Total
Number analyzed (Participants) | 197 | 196 | 393
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.4 (11.82) | 53.4 (11.11) | 52.4 (11.50)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 197 | 196 | 393
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 197 | 195 | 392
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 197 | 196 | 393
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 0 | 1
  Bulgaria | 18 | 18 | 36
  Hungary | 23 | 22 | 45
  Russia | 73 | 72 | 145
  Ukraine | 82 | 84 | 166
Weight [Mean (Standard Deviation); unit: kg] | 75.84 (16.884) | 74.93 (16.873) | 75.39 (16.863)
Height [Mean (Standard Deviation); unit: cm] | 162.6 (6.27) | 162.2 (6.67) | 162.4 (6.47)
Basal Metabolic Index [Mean (Standard Deviation); unit: kg/m2] | 28.72 (6.358) | 28.51 (6.197) | 28.62 (6.271)

OUTCOME MEASURES:

1. Primary Outcome: Duration in Days of Grade 4 Neutropenia in Chemotherapy Cycle 1
Description: Eligible subjects were randomized in a 1:1 ratio. Subjects were dosed with either the F 627 20 mg/dose PFS or Neulasta® 6 mg/dose as the study drug in each chemotherapy cycle. Subjects remained in their assigned treatment arm throughout the study. Subjects were dosed subcutaneously (SC) 24 to 28 hours after receiving TC chemotherapy (75 mg/m2 docetaxel + 600 mg/m2 cyclophosphamide) on Day 2 of each chemotherapy cycle that the subject underwent (up to 4 cycles). Grade 4 (severe) neutropenia was defined as ANC <0.5 × 109/L within the first 12 days of chemotherapy.
Time Frame: The first of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: ITT (Intent-to-Treat) population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 | Neulasta
Number analyzed (Participants) | 197 | 196
days | 0.2 (0.51) | 0.2 (0.45)

2. Secondary Outcome: Duration in Days of Use of Intravenous Antibiotic
Description: The duration of use of IV antibiotics was defined as the number of days in which IV antibiotics were administered
Time Frame: across all 4 chemotherapy cycles (average 84 days)
Population: ITT (Intent-to-Treat) population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 | Neulasta
Number analyzed (Participants) | 197 | 196
days | 0.3 (1.36) | 0.1 (0.70)

3. Secondary Outcome: Duration in Days of Hospitalization
Description: The duration in days of patients been hospitalized for febrile neutropenia (FN) or any infection. Febrile neutropenia is defined as a single oral temperature of ≥38.3°C (101°F) or a temperature of >38.0°C (100.4°F) sustained for >1 hour and ANC <0.5 x 10^9/L on the same day.
Time Frame: across all 4 chemotherapy cycles (average 84 days)
Population: ITT (Intent-to-Treat) population
Measure: Mean (Standard Deviation); unit: days
Arm/Group | F-627 | Neulasta
Number analyzed (Participants) | 197 | 196
days | 0.1 (0.78) | 0 (0.57)

4. Secondary Outcome: The Number of Participants With Grade 4 Neutropenia for Chemotherapy Cycle 1
Description: The number of participants with grade 4 neutropenia for chemotherapy cycle 1. Grade 4 (severe) neutropenia was defined as ANC <0.5 × 109/L within the first 12 days of chemotherapy.
Time Frame: The first of 4, 21-day chemotherapy cycles (average 3 weeks)
Population: ITT (Intent-to-Treat) population
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 | Neulasta
Number analyzed (Participants) | 197 | 196
Participants | 23 | 23

5. Secondary Outcome: The Number of Participants With Febrile Neutropenia Considering All Chemotherapy Cycles.
Description: The number of participants with febrile neutropenia, considering all chemotherapy cycles.
Time Frame: across all 4 chemotherapy cycles (average 84 days)
Population: ITT (Intent-to-Treat) population
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 | Neulasta
Number analyzed (Participants) | 197 | 196
Participants | 6 | 1

6. Secondary Outcome: The Number of Participants With Use of IV Antibiotics Considering All Chemotherapy Cycles.
Description: The number of participants with use of IV antibiotics, considering all chemotherapy cycles.
Time Frame: across all 4 chemotherapy cycles (average 84 days)
Population: ITT (Intent-to-Treat) population
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 | Neulasta
Number analyzed (Participants) | 197 | 196
Participants | 9 | 2

7. Secondary Outcome: The Number of Participants in Hospitalization for Febrile Neutropenia or Any Infection Considering All Chemotherapy Cycles
Description: The number of participants in hospitalization for febrile neutropenia or any infection, .
Time Frame: across all 4 chemotherapy cycles (average 84 days)
Population: ITT (Intent-to-Treat) population
Measure: Count of Participants; unit: Participants
Arm/Group | F-627 | Neulasta
Number analyzed (Participants) | 197 | 196
Participants | 1 | 1

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the time of randomization until end of treatment visit day 84 (total of 9 months).
Description: Treatment emergent AE was defined as any AE that began on or after study drug (F-627 or Neulasta) treatment up to the EOT visit or was a worsening of a pre-existing medical condition.
Arm/Group | F-627 | Neulasta
All-Cause Mortality (participants affected / at risk) | 1/197 | 2/196
Serious Adverse Events (participants affected / at risk) | 12/197 | 3/196
Other Adverse Events (participants affected / at risk) | 70/197 | 51/196
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | F-627 (N=197) | Neulasta (N=196)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
fatigue (General disorders) | 1 (1) | 0 (0)
diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
syncope (Nervous system disorders) | 1 (1) | 0 (0)
acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 1 (1) | 0 (0)
angioedema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Hepatitis toxic (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | F-627 (N=197) | Neulasta (N=196)
Bone pain (Musculoskeletal and connective tissue disorders) | 31 (54) | 23 (44)
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 (16) | 6 (9)
Leukocytosis (Blood and lymphatic system disorders) | 14 (58) | 10 (39)
Asthenia (Gastrointestinal disorders) | 13 (26) | 12 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/31/NCT03252431/Prot_000.pdf
  • Statistical Analysis Plan (2017-04-03): https://cdn.clinicaltrials.gov/large-docs/31/NCT03252431/SAP_001.pdf